CLINICAL TRIAL: NCT02561728
Title: Prospective Study to Evaluate Effectiveness of the Hanger Helmet vs the P Pod Helmet in Improving the Head and Face Symmetry
Brief Title: Hanger Helmet Study
Status: Withdrawn | Phase: Not Applicable | Type: Interventional
Why Stopped: No Participants Enrolled
Sponsor: Children's Hospital Medical Center, Cincinnati (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: 2015-1748
Record Dates: First submitted 2015-09-25; First posted 2015-09-28 (Estimated); Last update posted 2016-06-29 (Estimated); Status verified 2016-06

CONDITIONS: Plagiocephaly; Craniosynostosis
Keywords: Helmet; Hangar; P-Pod; Plagiocephaly; Surgery
MeSH Terms: conditions — Plagiocephaly; Craniosynostoses

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (2):
- Plagiocephaly (Experimental): Children with a misshaped head due to positioning. This is also known as flat head. Children with plagiocephaly will be treated with either the Hangar Helmet or the P-Pod helmet.
  Interventions: Device: Hangar Helmet; Device: P-Pod Helmet
- Craniosynostosis (Experimental): Craniosynostosis occurs when one or multiple sutures fuse too early. Several sutures may be fused alone or in combination. An open or endoscopic surgical procedure to open the suture(s) is necessary to allow for normal brain growth and development. After surgery a cranial remolding helmet is used to direct skull growth. Children with craniosynostosis will be treated with either the Hangar Helmet or the P-Pod helmet
  Interventions: Device: Hangar Helmet; Device: P-Pod Helmet

INTERVENTIONS:
Device: Hangar Helmet — Child will be fitted with the Hangar Helmet
Device: P-Pod Helmet — Child will be fitted with the P-Pod Helmet

SUMMARY:
The purpose of this study is to examine a group of patients requiring helmet therapy (either patients with plagiocephaly or post-surgical patients) to compare outcomes of infants treated with the Hanger helmet (Hanger, Inc.) to outcomes of infants treated with the P Pod Helmet (Lorica Scientific, LLC). Currently both helmets are prescribed at CCHMC. The investigators' goal is to determine which helmet is more effective in skull remodeling and to standardize the investigators' care for these patient types.

DETAILED DESCRIPTION:
The use of helmet therapy to correct abnormal head shape due to either positional plagiocephaly secondary to pressure on the posterior skull with infant position and furniture use or after minimally invasive surgery for craniosynostosis is currently the treatment of choice at Cincinnati Children's Hospital (CCHMC). Helmet treatment in children with positional plagiocephaly is initiated for infants between 4 and 9 months of age (at CCHMC). Helmet treatment for children undergoing surgery for craniosynostosis is initiated following endoscopic cranial vault and stip craniectomy surgery after swelling from the surgery has subsided (generally within two weeks of surgery). Treatment with helmet therapy has been shown to improve head shape in both patient diagnoses. There are two types of helmets available to the investigators' patients (Hanger Helmet and P Pod Helmet) and to date, no research has evaluated whether one helmet type is more efficient in reshaping the skull than the other type. The current study seeks to fill this gap in the literature by comparing the outcomes for infants treated with a Hanger Helmet to the outcomes for infants treated with a P Pod Helmet. The investigators will measure skull symmetry with a 3dMD camera and take routine cross lateral measurements with a caliper designed for this use. Infants participating in the study will be randomized using a computerized program, Minim.

ELIGIBILITY:
Inclusion Criteria:

* Diagnosis which requires helmet therapy treatment
* Under 10 months of age

Exclusion Criteria:

* Children who do not need helmet therapy

Max Age: 10 Months | Sex: All | Healthy Volunteers: No
Age Groups: Child
Enrollment: 0 (Actual)
Dates: Start 2016-07; Primary Completion 2022-10 (Estimated); Study Completion 2023-10 (Estimated)

PRIMARY OUTCOMES:
Root Mean Square (RMS) | 5 years
  RMA is measured by first taking a picture of the child's head with the helmet on with a 3dMD camera. RMS is a measurement unique to the 3dMD camera. RMS will be used to quantify symmetry by superimposing left and right quadrants and calculating the mean value of aggregate distances between surfaces.

CONTACTS AND LOCATIONS:
Overall Officials: John van Aalst, MD, Principal Investigator — Children's Hospital Medical Center, Cincinnati